CLINICAL TRIAL: NCT07193368
Title: Intra-Articular Polyacrylamide Hydrogel Injections Improve Pain and Function in Knee Osteoarthritis: A Multicenter Retrospective Study.
Brief Title: Intra-Articular Polyacrylamide Hydrogel Injections Improve Pain and Function in Knee Osteoarthritis
Acronym: HYDRO-KNEE
Status: Completed | Type: Observational
Sponsor: Feza Korkusuz MD (Other)
Collaborators: Dr. Özgür Oktay Nar Private Clinic, Bursa, Türkiye (Unknown); Contura International A/S, Copenhagen, Denmark (Unknown); Bursa City Hospital, Bursa, Türkiye (Unknown)
Responsible Party: Sponsor-Investigator, Feza Korkusuz MD, Feza Korkusuz, MD - Professor of Sports Medicine, Hacettepe University Faculty of Medicine, Hacettepe University
Organization: Hacettepe University (Other)
Other Study IDs: Approval No: 2025-14/3
Record Dates: First submitted 2025-09-12; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Knee Osteoarthritis; Osteoarthritis; Osteoarthritis of the Knee; Degenerative Joint Disease of the Knee
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — polyacrylamide gels; Injections, Intra-Articular

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Knee Osteoarthritis Patients: Patients diagnosed with knee osteoarthritis (Kellgren-Lawrence grade 2-4) who received a single intra-articular injection of 2.5% polyacrylamide hydrogel (Arthrosamid®, Contura, Denmark). Followed retrospectively for 12 months to assess pain (VAS) and function (WOMAC).
  Interventions: Biological: Polyacrylamide hydrogel 2.5% intra-articular injection

INTERVENTIONS:
Biological: Polyacrylamide hydrogel 2.5% intra-articular injection — A single intra-articular injection of 2.5% cross-linked polyacrylamide hydrogel (iPAAG), composed of 2.5% polyacrylamide and 97.5% non-pyrogenic water. The product (Arthrosamid®, Contura, Denmark) was administered under ultrasound guidance into the knee joint. Patients were followed retrospectively for 12 months to evaluate safety and effectiveness in reducing pain (VAS) and improving function (WOMAC).
  Other Names: Arthrosamid®; iPAAG injection

SUMMARY:
This study is designed to evaluate the effects of intra-articular injections of polyacrylamide hydrogel (Arthrosamid®) in patients with knee osteoarthritis. A total of 387 patients (593 knees) were treated across three medical centers in Türkiye.

The purpose of the study is to determine whether this injection can reduce knee pain and improve physical function in everyday life. Pain is being measured using a Visual Analogue Scale (VAS), and function is being assessed with the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 40 years
* Radiographic diagnosis of knee osteoarthritis (Kellgren-Lawrence grade 2-4)
* Received intra-articular 2.5% polyacrylamide hydrogel injection

Exclusion Criteria:

* Prior knee surgery before PAAG injection
* Malignancy, local infection, or septic arthritis
* Inflammatory joint disease (e.g., rheumatoid arthritis)
* Pregnancy
* Avascular necrosis
* Advanced varus or valgus knee deformity

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 40 years and older diagnosed with knee osteoarthritis (KL grade 2-4) who were treated with a single intra-articular polyacrylamide hydrogel injection at three medical centers in Türkiye and followed retrospectively for 12 months.
Sampling Method: Non-Probability Sample
Enrollment: 387 (Actual)
Dates: Start 2023-02-11 (Actual); Primary Completion 2025-06-24 (Actual); Study Completion 2025-06-24 (Actual)

PRIMARY OUTCOMES:
Change in Knee Pain (VAS Score) | Baseline and 12 months after injection
  Pain intensity will be measured using the Visual Analogue Scale (VAS; 0-10, with 0 = no pain and 10 = worst pain). Baseline values will be compared with values at 12 months after injection.
Change in Physical Function (WOMAC Function Subscale) | Baseline and 12 months after injection
  Physical function will be assessed using the WOMAC Function subscale (0-68; higher scores indicate worse function). Baseline values will be compared with values at 12 months after injection.
Change in Total WOMAC Score | Baseline and 12 months after injection
  Overall knee function and symptoms will be assessed using the WOMAC total score (0-100; higher scores indicate worse symptoms and function). Baseline values will be compared with values at 12 months after injection.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Faculty of Medicine, Department of Sports Medicine, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No